CLINICAL TRIAL: NCT00655421
Title: Comparing the Test Characteristics of Three Oral Cancer Screening Techniques:1)Unaided Visual Examination 2)VelScope Examination and 3)Toluidine Blue Application, by Trained Primary Health Care Workers in Mumbai, India.
Brief Title: Oral Cancer Screening in Mumbai, India by Primary Health Care Workers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: American Cancer Society, Inc. (Other); Emory University (Other)
Responsible Party: Dr.S.S.Shastri/Professor and Head, Department,Preventive Oncology, Tata Memorial Hospital, Mumbai, India
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 391
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Oral Cancer; Precancerous Conditions
Keywords: screening; oral precancers; tobacco users; VELScope; Visual Inspection; Toluidine Blue
MeSH Terms: conditions — Mouth Neoplasms; Precancerous Conditions; Tobacco Use

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Unaided (Experimental): Unaided Visual Inspection of the Oral Cavity
  Interventions: Other: Unaided Visual Inspection
- VelScope (Experimental): VelScope assisted examination of the oral cavity
  Interventions: Device: VelScope
- Toluidine (Experimental): Examination of oral cavity after the local application of Toluidine Blue dye
  Interventions: Other: Toluidine Blue Assisted Oral Examination

INTERVENTIONS:
Other: Unaided Visual Inspection — Simple unaided visual inspection of the oral cavity with a bright white light source by trained Primary Health Care Worker
  Arms: Unaided
Device: VelScope — Examination of the oral cavity through a VelScope by trained Primary Health Care Worker
  Arms: VelScope
Other: Toluidine Blue Assisted Oral Examination — Examination of the oral cavity after the local application of Toluidine Blue dye by trained Primary Health Care Worker
  Arms: Toluidine

SUMMARY:
A feasibility study to compare the test characteristics of three different oral cancer screening techniques performed by trained primary health care workers:1)Unaided Visual Inspection, 2)VelScope Assisted Examination, and 3) Examination after application of Toluidine Blue dye.

DETAILED DESCRIPTION:
Oral cancer is the most common cancer among men in India mainly due to the habit of using smokeless tobacco. Pre-cancerous lesions like leukoplakia, melanoplakia, erythroplakia,oral submucous fibrosis and indolent ulcers can be easily detected by periodic examination of the oral cavity of the at-risk populations. Several methods of oral cancer screening have been tried over the past three-four decades with varying success. This study investigates the feasibility of application and compares the test characteristics of three oral cancer screening techniques: Unaided Visual Inspection, VelScope assisted examination and examination after application of Toluidine blue dye by primary health care workers among tobacco users attending a cancer early detection clinic, in Mumbai, India.

ELIGIBILITY:
Inclusion Criteria:

* The study participants will be apparently healthy males with tobacco habit ( present tobacco users and those who have quit within past six months),
* above 18 years of age,
* attending Preventive Oncology clinic.

Exclusion Criteria:

* Participants with frank oral cancers will not be recruited in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility and efficacy of performance of the three oral cancer screening tests viz. naked eye unaided examination , examination using VELScope and after application of Toluidine Blue by trained primary health workers. | six months

SECONDARY OUTCOMES:
To estimate the test characteristics of each of the three oral cancer screening techniques. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Surendra S Shastri, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- See also: Customized optical device helps dentists to detect oral cancer — http://www.medicalnewstoday.com